CLINICAL TRIAL: NCT05621616
Title: A Phase 3, Open Label, Multicenter, Baseline-Controlled Sequential Dose Titration Study Followed by a Fixed Dose Observation Period to Evaluate Pharmacokinetics, Efficacy and Safety of Mirabegron Prolonged-Release Microgranula-Based Suspension in Children From 6 Months to Less Than 3 Years of Age With Neurogenic Detrusor Overactivity
Brief Title: A Study to Learn How Effective and Safe the Drug 'Mirabegron' is and How Long it Stays in the Body of Children Aged 6 Months to Less Than 3 Years of Age With Neurogenic Detrusor Overactivity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 178-CL-207; 2021-005455-37 (EudraCT Number); 2023-507903-74 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Neurogenic Detrusor Overactivity
Keywords: Neurogenic Detrusor Overactivity; Pediatric acceptability; Bladder capacity; Pharmacokinetics of mirabegron
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mirabegron (Experimental): Participants will receive mirabegron prolonged-release microgranula-based oral suspension.
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — Participants will receive mirabegron prolonged-release microgranula-based oral suspension once daily. The initial dose of mirabegron will be based on the participant's weight.
  The initial low dose will be up-titrated to a higher dose at weeks 2, 4 or 8 unless the participant is determined to be effectively treated with the low dose, based on urodynamics and the participants'e-diary.
  Other Names: Betanis; Betmiga; Myrbetriq; YM178

SUMMARY:
People with neurogenic detrusor overactivity (NDO) have poor bladder control because of how their nerves to the bladder are wired. This can cause high pressure in the bladder, causing it to leak urine by accident (incontinence). Mirabegron has already been approved for adults with bladder problems and for children 3 years and older. This study will learn if mirabegron can help young children with NDO. The children will be from 6 months to up to 3 years old.

The main aim of this study is to learn if mirabegron increases how much urine the bladder holds (maximum cystometric capacity, or Maximum Cystometric Capacity [MCC]) in young children with NDO. An increase in MCC will prevent high pressure in the bladder.

Children from 6 months to up to 3 years old who have NDO can take part. They must weigh 9 kilograms (kg) or more. They will already be fitted with a tube (catheter) in their bladder. They will use this to drain urine from their bladder regularly during the day. This is called clean intermittent catheterization (CIC).

There will be 2 groups in the study. Young children who aren't taking certain medicines for NDO will be in group A. Young children who are taking certain medicines for NDO will be in group B. Children in group B will stop taking these medicines before they start taking mirabegron. Treatment in group B will be delayed to allow the medicines to be cleared from the body before they start taking mirabegron. Both groups (A and B) will have the same treatment and dose of mirabegron and will have the same checks throughout the study.

Mirabegron will be squirted from a syringe into the children's mouths, followed by a sip of water. This will happen once a day for up to 52 weeks (1 year). They will start on a low dose, adjusted for their weight. The dose may be increased to a higher dose if the study doctor thinks the child will benefit from the higher dose.

Children will have safety checks throughout the study. Other tests will include checking how the bladder fills and empties plus an ultrasound of the bladder area.

There will be several clinic visits during the study. There will be fewer clinic visits if a child stays on the low dose of mirabegron. Then, the clinic will phone the caregiver about 1 month after the last dose of mirabegron to check if there are any further medical problems.

ELIGIBILITY:
Inclusion Criteria:

* Participant's weight is a minimum of 9 kg.
* Participant has a previous myelomeningocele (documented at the screening visit).
* Participant has a diagnosis of neurogenic detrusor overactivity (NDO) confirmed by urodynamic investigation at baseline (day 1). The diagnosis of NDO should be confirmed by the presence of ≥ 1 involuntary detrusor contraction > 15 cm H2O from baseline detrusor pressure, and/or a decrease in bladder compliance leading to an increase in baseline detrusor pressure of > 20 cm H2O.
* Participant has a diagnosis of detrusor sphincter dyssynergia (DSD).
* Participant is using clean intermittent catheterization (CIC).
* Participant is suitable for a regimen of 4 to 6 CICs per day, fixed for the duration of the study using the 7-day baseline e-diary.
* Participant is able to swallow the study drug.
* Participant's legally authorized representative (LAR) is willing and able to comply with the study requirements (including compliant use of the e-diary) and with the concomitant medication restrictions.
* Participant's LAR agree not to allow participant to participate in another interventional study while receiving study intervention and throughout the pretreatment period.

Exclusion Criteria:

* Participant has a bladder capacity less than 25% of expected age-related capacity, confirmed by urodynamic investigation at baseline (day 1).
* Participant has vesicoureteral reflux grade 3 to 5.
* Participant has a known genitourinary condition, other than NDO, that may cause overactive contractions and/or incontinence (e.g., bladder exstrophy, urinary tract obstruction, urethral diverticulum or fistula) or kidney/bladder stones or another persistent local pathology that may cause urinary symptoms.
* Participant has had an indwelling urinary catheter within 4 weeks prior to the baseline visit.
* Participant has undergone bladder augmentation surgery.
* Participant with surgically corrected underactive sphincter.
* Participant receives electrostimulation therapy, if started within 30 days before visit 1 screening or is expected to start during the study period. Participants who are on an established regimen (defined as starting more than 30 days before visit 1 screening) may remain on this for the duration of the study.
* Participant has been administered intravesical botulinum toxin; except if given > 4 months prior to visit 1 screening and the participant experiences symptoms comparable to those existing prior to the botulinum toxin injections.
* Participant has a current symptomatic urinary tract infection (UTI) confirmed by urinalysis (urine culture containing > 100,000 cfu/mL) at baseline. If at screening and start of washout a UTI is present, the participant will be eligible for enrollment if the UTI has been treated successfully prior to baseline. If a symptomatic UTI is present at baseline, all baseline assessments should be postponed for a maximum of 7 days until the UTI is successfully treated. Successful treatment is defined as a symptom free patient with a white blood cell count in the urine < 100/microliter and urine culture below 100,000 cfu/mL.
* Participant is using prohibited medications.
* Participant has a diagnosis of central or congenital nephrogenic diabetes insipidus.
* Participant with severe gastrointestinal (GI) condition (including toxic megacolon) or any of the following GI conditions: partial or complete obstruction, decreased motility like paralytic ileus or at risk for gastric retention.
* Participant suffers from malnutrition or is severely overweight.
* Participant has an average QT interval corrected by Bazett's formula (QTcB) > 440 ms (based on the QTcB mean from the screening and baseline ECG triplicates), history of QTc prolongation or risk of QT prolongation (e.g., hypokalemia, Long QT Syndrome (LQTS), or family history of LQTS, exercise induced syncope).
* Participant has severe renal impairment (estimated glomerular filtration rate (eGFR) < 30 mL/min per 1.73 m^2 for participants 1 year of age and older; serum creatinine ≥ 2 × ULN, with ULN defined as 97.5th percentile for participants 6 to < 12 months of age.).
* Participant's aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is ≥ 2 × upper limit of normal (ULN) or total bilirubin (TBL) greater than or equal to 1.5 × ULN.
* Participant has a current or previous history of epilepsy.
* Participant has a history or presence of any malignancy prior to visit 1 screening.
* Participant has any other clinically significant out of range results of urinalysis, biochemistry, hematology or coagulation.
* Participant has an established hypertension and systolic or diastolic blood pressure greater than the 99th percentile of their normal range determined by gender, body size and age, plus 5 mmHg.
* Participant has a (median) resting heart rate > 99th percentile.
* Participant has any clinically significant or unstable medical condition or disorder which precludes the participant from participating in the study.
* Participant has known or suspected hypersensitivity to mirabegron, any of the excipients used in the current formulation or previous severe hypersensitivity to any drug.
* Participant has participated in another clinical trial and/or has taken an investigational drug within 30 days (or 5 half-lives of the drug, or the limit set by national law, whichever is longer) prior to visit 1 screening.
* Participant is being breast-fed by a woman taking any prohibited medication or fed with a milk product in which the presence of prohibited medication ingredients cannot be excluded.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Week 24 in Maximum Cystometric Capacity (MCC) | Baseline and week 24
  MCC is maximum bladder capacity reached at end of filling cytometry.

SECONDARY OUTCOMES:
Change from baseline in bladder compliance | Baseline and weeks 4 and 24
  Bladder compliance is calculated by change in volume divided by change in pressure during filling of the bladder.
Change from baseline in filling volume until first detrusor contraction (>15cm H2O) | Baseline and weeks 4 and 24
  Change in bladder volume calculated by urodynamic assessments.
Change from baseline in number of uninhibited detrusor contractions until leakage or until maximum 135% of age-related bladder capacity | Baseline and weeks 4 and 24
  Change in number of of uninhibited detrusor contractions is calculated by urodynamic assessments.
Change from baseline in maximum catheterized daytime volume | Baseline and up to week 52
  Based on participant e-diary.
Change from baseline in average catheterized daytime volume | Baseline and up to week 52
  Based on participant e-diary.
Change from baseline in average morning catheterized volume | Baseline and up to week 52
  E-diary measure based on first catheterization after participant wakes up.
Change from baseline in number of leakage episodes per 24 hours | Baseline and up to week 52
  Based on participant e-diary.
Change from baseline in number of dry days per 7 days | Baseline and up to week 52
  Based on participant e-diary, dry defined as leakage-free.
Acceptability by pediatric oral medicine acceptability questionnaire for caregivers (P-OMAQ-C) | Baseline and weeks 4, 24 and 52
  The P-OMAQ-C uses a 5-point numerical rate scale to measure acceptability of use of the tablet formulation with questions related to taste, smell and administration of study medication. Acceptability questionnaires to be completed by caregivers on an electronic device.
Frequency of adverse events (AE) | Up to week 54
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator and events related to the (study) procedures.
Number of Participants With Vital Sign Abnormalities and/or AEs | Up to week 54
  Number of participants with potentially clinically significant vital sign values.
Number of participants with laboratory value abnormalities and/or AEs | Up to week 52
  Number of participants with potentially clinically significant laboratory values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to week 54
  Number of participants with potentially clinically significant ECG values.
Number of participants with upper urinary tract ultrasound abnormalities and/or AEs | Up to week 52
  Number of participants with potentially clinically significant upper urinary tract ultrasounds.
PK of mirabegron in plasma: Area under the concentration-time curve per 24 hours (AUC24) | Up to week 52
  AUC24 will be recorded from the PK plasma samples collected.
PK of mirabegron in plasma: Concentration immediately prior to dosing (Ctrough) | Up to week 52
  Ctrough will be recorded from the PK plasma samples collected.
PK of mirabegron in plasma: Apparent clearance (CL/F) | Up to week 52
  CL/F will be recorded from the PK plasma samples collected.
PK of mirabegron in plasma: Apparent volume of distribution (VzF) | Up to week 52
  VzF will be recorded from the PK plasma samples collected.
PK of mirabegron in plasma: Maximum concentration (Cmax) | Up to week 52
  Cmax will be recorded from the PK plasma samples collected.
PK of mirabegron in plasma: Time of maximum concentration (Tmax) | Up to week 52
  Tmax will be recorded from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (4):
- Site DE49002, Hanover, Germany
- Philippines (2):
  - Site PH63001, Quezon
  - Site PH63002, Quezon City
- Site PL48001, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.